CLINICAL TRIAL: NCT02957630
Title: A Single Center, Randomized,Open-label,Controlled, Three-arm Study to Evaluate the Effect of a New Combined Oral Contraceptive (COC) Containing 15 mg Estetrol (E4) and 3 mg Drospirenone (DRSP) and of Two Reference COCs Containing Either 30 mcg Ethinylestradiol (EE) and 150 mcg Levonorgestrel (LNG) or 20 mcg EE and 3 mg DRSP on Endocrine Function, Metabolic Control and Hemostasis During 6 Treatment Cycles
Brief Title: "E4/DRSP Endocrine Function, Metabolic Control and Hemostasis Study"
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Estetra (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MIT-Es0001-C201; 2016-001316-37 (EudraCT Number)
Record Dates: First submitted 2016-10-25; First posted 2016-11-08 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2017-03

CONDITIONS: Contraception; Liver Metabolism; Hemostasis Parameter
Keywords: Estetrol (E4); Drospirenone (DRSP); Ethinylestradiol (EE); Levonorgestrel (LNG); Oral contraceptive; Prevention of pregnancy; Hemostasis; Metabolism
MeSH Terms: interventions — Estetrol; drospirenone; Ethinyl Estradiol; Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 15 mg E4/3 mg DRSP (Experimental): 15 mg estetrol/3 mg drospirenone combined oral contraceptive
  Interventions: Drug: 15 mg E4/3 mg DRSP
- 30 mcg EE/150 mcg LNG (Active Comparator): 30 mcg ethinylestradiol/150 mcg levonorgestrel combined oral contraceptive
  Interventions: Drug: 30 mcg EE/150 mcg LNG
- 20 mcg EE/3 mg DRSP (Active Comparator): 20 mcg ethinylestradiol/3 mg drospirenone combined oral contraceptive
  Interventions: Drug: 20 mcg EE/3 mg DRSP

INTERVENTIONS:
Drug: 15 mg E4/3 mg DRSP — 15 mg E4 combined with 3 mg DRSP administered in a 24/4-day regimen (i.e. 24 days of pink active tablets followed by 4 days of white placebo tablets). One tablet per day orally for 6 treatment cycles.
  Other Names: 15 mg estetrol and 3 mg drospirenone
  Arms: 15 mg E4/3 mg DRSP
Drug: 30 mcg EE/150 mcg LNG — 30 mcg EE combined with 150 mcg LNG administered in a 21/7-day regimen (i.e. 21 days of yellow active tablets followed by 7 days of white placebo tablets). One tablet per day orally for 6 treatment cycles.
  Other Names: 30 mcg ethinylestradiol and 150 mcg levonorgestrel
  Arms: 30 mcg EE/150 mcg LNG
Drug: 20 mcg EE/3 mg DRSP — 20 mcg EE combined with 3 mg DRSP administered in a 24/4-day regimen (i.e. 24 days of pink active tablets followed by 4 days of white placebo tablets). One tablet per day orally for 6 treatment cycles.
  Other Names: 20 mcg ethinylestradiol and 3 mg drospirenone
  Arms: 20 mcg EE/3 mg DRSP

SUMMARY:
The proposed study will provide an assessment of the effect of this combination on endocrine function, metabolic control and hemostasis during 6 treatment cycles. This will be compared to the effects of two reference COCs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult woman
* Negative pregnancy test at subject screening and randomization
* Aged 18-50 years (inclusive) at the time of signing the ICF
* Good physical and mental health on the basis of medical, surgical and gynecological history, physical examination, gynecological examination, clinical laboratory, ECG, echocardiography and vital signs
* BMI from 18.0 to 30.0 kg/m², inclusive, at time of screening visit
* Able to fulfil the requirements of the protocol and have indicated a willingness to participate in the study by providing written informed consent

Exclusion Criteria:

* Known hypersensitivity to any of the investigational product ingredients
* Smoking if > 35 years old
* Dyslipoproteinemia or use of antilipidemic agent
* Known diabetes mellitus
* Current use of antidiabetic drugs, including insulin
* Arterial hypertension
* Any condition associated with an increased risk of venous thromboembolism and/or arterial thromboembolism.
* Any condition associated with abnormal uterine/vaginal bleeding.
* Presence of an undiagnosed breast mass
* Current symptomatic gallbladder disease
* History of pregnancy- or COC-related cholestasis
* Presence or history of severe hepatic disease
* Presence or history of pancreatitis if associated with hypertriglyceridemia
* Porphyria
* Presence or history of benign liver tumors (focal nodular hyperplasia and hepatocellular adenoma)
* Presence of renal impairment (glomerular filtration rate [GFR] <60 mL/min/1.73m²)
* Hyperkalemia or presence of conditions that predispose to hyperkalemia
* Presence or history of hormone-related malignancy
* History of non-hormone-related malignancy within 5 years before screening; subjects with a non-melanoma skin cancer are allowed in the study
* Use of drugs potentially triggering interactions with COCs
* History of alcohol or drug abuse within 12 months prior to screening
* Presence or history of thyroid disorders
* Participation in another investigational drug clinical study within 1 month (30 days) or have received an investigational drug within the last 3 months (90 days) prior to randomization. Subjects who participated in an oral contraceptive clinical study using Food and Drug Administration (FDA)/European Union (EU) approved active ingredients, may be randomized 2 months (60 days) after completing the preceding study
* Sponsor, contract research organization (CRO) or Principal Investigator's (PI's) site personnel directly affiliated with this study
* Is judged by the PI to be unsuitable for any reason

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2016-09; Primary Completion 2017-10-09 (Actual); Study Completion 2017-10-09 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of prothrombin fragment 1+2 | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Plasma concentration of APC resistance (ETP-based, APTT-based) | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Plasma concentration of D-dimer | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Plasma concentration of factor VII | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Plasma concentration of factor VIII | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Plasma concentration of von Willebrand factor | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Plasma concentration of factor II | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Plasma concentration of antithrombin | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Plasma concentration of free and total Protein S | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Plasma concentration of protein C | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Plasma concentration of plasminogen activator inhibitor type-1 (PAI-1) | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Plasma concentration of tissue type plasminogen activator (t-PA) | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Plasma concentration of plasminogen | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Plasma concentration of free tissue factor pathway inhibitor (TPFI) | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Plasma concentration of E-selectin | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Plasma concentration of fibrinogen | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of insulin | At screening, between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of glucose | At screening, between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of C-peptide | At screening, between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for Cycles 3 and 6 (1 cycle = 28 days).
Plasma concentration of glycated hemoglobin (HbA1c) | At screening, between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Homeostasis Model Assessment - Insulin Resistance (HOMA-IR) | At screening, between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Oral glucose tolerance test (OGTT) | At 0 (pre-glucose challenge), 30, 60, 90, 120 and 180 minutes after glucose challenge during pretreatment Cycle; at 0 (pre-glucose challenge), 30, 60, 90, 120 and 180 minutes after glucose challenge during Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of prolactin | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of follicle-stimulating hormone (FSH) | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of luteinizing hormone (LH) | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of estradiol (E2) | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of progesterone (P) | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of thyroïd stimulating hormone (TSH) | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of free thyroxine (fT3)/free triiodothyronine (fT4) | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of dihydroepiandrostenedione (DHEAS) | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of androstenedione | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of total testosterone (T) | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of dihydrotestosterone (DHT) | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of total cortisol | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of aldosterone | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of high density lipoprotein (HDL)-cholesterol | At screening, between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of low density lipoprotein (LDL)-cholesterol | At screening, between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of total cholesterol | At screening, between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of triglycerides | At screening, between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of lipoprotein (a) | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of apoliporotein A1 | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of apoliporotein B | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of C-reactive protein | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of corticosteroid binding globulin (CBG) | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of sex hormone binding globulin (SHBG) | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of thyroxin binding globulin (TBG) | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).
Serum concentration of angiotensinogen | Between Days 18 and 21 for the pretreatment Cycle, and between Days 18 and 21 for the Cycles 3 and 6 (1 cycle = 28 days).

SECONDARY OUTCOMES:
Number of subjects with adverse events as a measure of safety and tolerability | From up to 28 days before randomization to maximum Day 4 of the Cycle 7 (1 cycle = 28 days).
Serum concentration of lactate dehydrogenase (LDH) 1 and 2 | Between Days 18 and 21 for the pretreatment Cycle and between Days 18 and 21 for the Cycle 6 (1 cycle = 28 days)
Serum concentration of tropinin T and I | Between Days 18 and 21 for the pretreatment Cycle and between Days 18 and 21 for the Cycle 6 (1 cycle = 28 days)
Electrocardiogram (ECG) parameters | At screening and between Days 18 and 21 for Cycle 6 (1 cycle = 28 days).
  The following ECG parameters will be recorded: heart rate, PR-interval, QRS-duration, QT-interval, QTc interval (Fridericias's)
Echocardiographic parameters | At screening and between Days 18 and 21 for Cycle 6 (1 cycle = 28 days).
Change from baseline to end of treatment in the different items of the menstrual distress questionnaires (MDQ) form C | At pretreatment Cycle and between Days 18 and 21 for Cycle 6 (1 cycle = 28 days).

CONTACTS AND LOCATIONS:
Overall Officials: Christine Klipping, Principal Investigator — Dinox BV
Locations (1):
- Dinox BV, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided